CLINICAL TRIAL: NCT06549751
Title: A Phase 1 Study Of Patient-Derived Multi-Tumor-Associated Antigen Specific T Cells (MT-601) Administered To Patients With Locally Advanced Unresectable or Metastatic Pancreatic Cancer
Brief Title: MT-601 Administered To Patients With Locally Advanced Unresectable or Metastatic Pancreatic Cancer
Acronym: PANACEA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marker Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MRKR-22-601-02
Record Dates: First submitted 2024-06-06; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation (Experimental): Cohort -1 / 100 million cells / 3-6 patients Cohort 1 / 200 million cells / 3-6 patients Cohort 1 / 400 million cells / 3-6 patients
  Interventions: Biological: MT-601
- Expansion (Experimental): The Dose Expansion portion will begin after completion of the Dose Escalation portion and focus on the efficacy of MT-601 as add-on to front-line chemotherapy. The dose level for the expansion portion of the study will be selected based on totality of the data. The primary objective is to evaluate clinical efficacy for the dose expansion. A total of 20 to 25 patients are planned to be enrolled.
  Interventions: Biological: MT-601

INTERVENTIONS:
Biological: MT-601 — Cellular Therapy

SUMMARY:
The goal of this clinical trial is to assess safety and tolerability of escalating doses of MT-601 administered during the off week of chemotherapy regimen for patients with pancreatic cancer. The main question[s] it aims to answer are: safety and efficacy • overall response rate and duration of response. Participants will meet all applicable inclusion criteria prior to chemotherapy and must agree to provide apheresis material.

DETAILED DESCRIPTION:
The Dose Escalation portions will proceed using a standard 3+3 design. Flat doses of MT-601 will be administered ranging from 200 million cells to 400 million cells. For the Dose Expansion, MT-601 will be administered at the dose determined to be safe based on the results from the Dose Escalation portion. Front-line chemotherapy (FOLFIRINOX or gemcitabine/nab-paclitaxel) will be administered as per standard of care. MT-601 will be administered intravenously over 10 minutes (± 5 minutes) during the "off" week of front-line chemotherapy. Patients will receive up to 6 infusions of MT-601 approximately every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed newly diagnosed locally advanced, unresectable or metastatic pancreatic adenocarcinoma (excluding other pancreatic malignancies such as acinar cell carcinomas or neuroendocrine cell neoplasms, etc.).
2. Eligible for reassessment following 2 months of front-line chemotherapy (FOLFIRINOX or gemcitabine/nab-paclitaxel): Patient must have experienced a response of SD, PR, or CR per RECIST v1.1 after 2 months of front-line chemotherapy (FOLFIRINOX or gemcitabine/nab-paclitaxel).
3. ≥18 years of age prior to administration of MT-601.
4. Measurable or evaluable disease per RECIST v1.1 at the time of screening.
5. Must have sufficient leukapheresis material to manufacture autologous MT601.
6. Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
7. Life expectancy ≥12 weeks.
8. Pulse oximetry of >90% on room air in patients with previous radiation therapy.
9. Adequate organ function, as defined below:

   * Absolute neutrophil count (ANC) ≥1.5 × 109/L
   * Platelets ≥75 × 109/L
   * Hemoglobin ≥9 g/dL (can be transfused)
   * International normalized ratio (INR) or prothrombin time (PT) ≤1.5 × upper limit of normal (ULN) (unless patient receiving stable dose of anticoagulant therapy as long as PT or INR in therapeutic range of intended anticoagulant)
   * Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) PTT or aPTT ≤ 5 seconds above ULN (unless patient receiving stable dose of anticoagulant therapy "a" as long as PT or INR in therapeutic range of intended anticoagulant)
   * Total bilirubin ≤2 × ULN
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN OR ≤5 × ULN if liver has tumor involvement
   * Serum creatinine OR calculated (as per institutional standards) creatinine clearance ≤2 × ULN OR measured or calculated ≥50 mL/min for patients "a" If receiving anticoagulation, the patient must have no active bleeding within 14 days prior to baseline assessment.
10. Sexually active patients must be willing to utilize one of the highly effective birth control methods or practice complete abstinence between initiation of screening for MT-601 infusion and 6 months after the last MT-601 infusion. Male patients who are sexually active must agree to use a condom during this period.
11. Disease imaging prior to administration of front-line chemotherapy and reimaging prior to administration of MT-601.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
During Dose Escalation - assess the safety and tolerability of escalating doses of MT-601 administered during the off week of chemotherapy regimen. | Through study completion. Approximately 3 years
  * Dose-limiting toxicities (DLTs)
  * Safety (including but not limited to): treatment-emergent adverse events, SAEs, deaths, and clinical laboratory abnormalities per NCI CTCAE, Version 5.0
During Dose Expansion - estimate overall response rate (ORR) of MT-601 | Through study completion. Approximately 3 years
  To estimate overall response rate (ORR) of MT-601 administered during the off week of chemotherapy regimen (RECIST v1.1) ORR to be measured by disease assessments conducted prior to treatment, at baseline, 8 weeks, 16 weeks and during active follow-up visits which will occur every 8 weeks (starting from Week 24), using RECIST v1.1
During Dose Expansion - estimate duration of response (DOR) of MT-601 | Through study completion. Approximately 3 years
  To estimate duration of response (DOR)of MT-601 administered during the off week of chemotherapy regimen (RECIST v1.1) DRR to be measured by disease assessments conducted prior to treatment, at baseline, 8 weeks, 16 weeks and during active follow-up visits which will occur every 8 weeks (starting from Week 24), using RECIST v1.1

SECONDARY OUTCOMES:
During Dose Escalation and Dose Expansion - determine the Efficacy of MT-601 | Through study completion. Approximately 3 years
  To assess anti-tumor activity of MT-601 administered during the off week of chemotherapy regimen based on RECIST v1.1 and overall survival (OS)
  * ORR and DOR
  * Disease control rate (DCR), time to response (TTR), PFS
  * OS
During Dose Expansion - assess safety and tolerability of MT-601 | Through study completion. Approximately 3 years
  To assess safety and tolerability of MT-601 administered during the off week of chemotherapy regimen
  -Safety (including but not limited to): TEAEs, SAEs, deaths, and clinical laboratory abnormalities per NCI CTCAE Version 5.0

OTHER OUTCOMES:
Exploratory: During Dose Escalation and Dose Expansion - examine the expansion, persistence, clonality and anti-tumor immune effects of the adoptively transferred, autologous MT-601, as well as the presence of epitope spreading in all groups | Through study completion. Approximately 3 years
  * Explore markers of immune function, cell targeting, signaling pathways and disease status
  * Examine ORR, DOR, DCR, TTR, and PFS based on iRECIST
Exploratory: During Dose Escalation and Dose Expansion - assess anti-tumor activity of MT-601 administered during the off week of chemotherapy regimen based on iRECIST | Through study completion. Approximately 3 years
  * Explore markers of immune function, cell targeting, signaling pathways and disease status
  * Examine ORR, DOR, DCR, TTR, and PFS based on iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Allison, BS, Study Director — Marker Therapeutics

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be developed if it is decided that the results of this study may be published or presented at scientific meetings.